CLINICAL TRIAL: NCT04039373
Title: An Open-label, Single-sequence Study to Investigate the Effects of BMS-986256 at Steady State on the Single Dose Pharmacokinetics of Mycophenolate Mofetil in Healthy Male Participants
Brief Title: Effects of BMS-986256 at Steady State on the Single Dose Pharmacokinetics of Mycophenolate Mofetil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IM026-022
Record Dates: First submitted 2019-07-22; First posted 2019-07-31 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: BMS-986256; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: BMS-986256 — specified dose on specified days
Drug: Mycophenolate Mofetil — specified dose on specified days

SUMMARY:
A Study to Investigate BMS-986256 at steady state and its effect on Mycophenolate Mofetil exposure in Healthy Male Participants

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant, defined as having no clinically significant active or ongoing medical condition, physical examination abnormality, abnormal ECG finding, with no current use of tobacco
* A negative QuantiFERON-TB Gold® test result at screening or documentation of a negative result within 3 months of the screening visit and a weight ≥ 50 kg and BMI between 18.0 and 32.0 kg/m2 inclusive at screening.
* Participants must not be current users (within 6 months before screening) of tobacco or tobacco- or nicotine-containing products; they must also be willing to refrain from using any of these products during their participation in the study.
* Men who are sexually active with women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception (APPENDIX 4) for the duration of treatment with BMS-986256 or MMF, plus 5 half-lives of BMS-986256 (19 days) plus an additional 90 days (duration of sperm turnover) for a total of 109 days post treatment. In addition, participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Any significant acute or chronic medical illness or condition, in the opinion of the investigator in addition to prior exposure to BMS-986256
* Major surgery within 4 weeks before study treatment administration, drug abuse or drug addiction.
* Participants who have smoked or used smoking cessation or other nicotine-containing products within 6 months before the first dose of study drug.
* History or presence of malignancy including hematological malignancies. However,participants with a history of basal cell or squamous cell carcinoma of the skin that has been completely and successfully treated with no evidence of recurrence may not be excluded, at the discretion of the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Mycophenolic Acid (MPA) PK parameter: Maximum observed plasma concentration (Cmax) | days 1-5 and days 26 -30
mycophenolic acid (MPA) PK parameter: area under the concentration-time curve from time zero to the time of the last quantifiable concentration AUC (0-T) | Days 1-5 and Days 26 -30
Mycophenolic Acid (MPA) PK parameter:area under the concentration-time curve from time zero extrapolated to infinite time AUC (INF) | Days 1-5 and days 26 -30

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | up to 51 days
Incidence of Serious Adverse Events (SAEs) | up to 51 days
Number of Clinically significant changes in lab assessment of blood serum | up to 51 days
Number of Clinically significant changes in assessment of blood | up to 51 days
Number of Clinically significant changes in lab assessment of urine | up to 51 days
Vital signs of blood pressure | up to 51 days
Vital signs of body temperature | up to 51 days
Vital signs of respiratory rate | up to 51 days
Number of Participants with abnormal physical examination findings | up to 51 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm